CLINICAL TRIAL: NCT03003988
Title: Effects of 28 Days of Different Forms of Creatine Supplementation on Muscle Creatine, Body Composition and Exercise Performance in Recreationally Active Males
Brief Title: Physiological Effects of Creatine Supplementation in Active Males
Acronym: NB4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Nutrabolt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB2014-0503FX
Record Dates: First submitted 2016-12-14; First posted 2016-12-28 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Dietary Supplementation
MeSH Terms: interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Creatine monohydrate (Experimental): Creatine monohydrate (6.0 g.) + dextrose (0.5 g.)
  Interventions: Dietary Supplement: Creatine monohydrate
- Creatine nitrate (Active Comparator): Creatine nitrate (5.0 g. creatine monohydrate + 1.5 g. creatine nitrate that provides 1.0 g. of creatine and 0.5 g. nitrate in 2:1 ratio).
  Interventions: Dietary Supplement: Creatine nitrate
- Placebo (Placebo Comparator): 6.5 g. dextrose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine monohydrate — Creatine monohydrate (6.0 g) + dextrose (0.5 g)
  Arms: Creatine monohydrate
Dietary Supplement: Creatine nitrate — Creatine nitrate (5.0 g creatine monohydrate + 1.5 g. creatine nitrate that provides 1.0 g. of creatine and 0.5 g. nitrate in 2:1 ratio)
  Arms: Creatine nitrate
Dietary Supplement: Placebo — Placebo (6.5 g dextrose)
  Arms: Placebo

SUMMARY:
This study was designed to examine how different forms of creatine impact active males.

DETAILED DESCRIPTION:
This study examined the effects of different formulations of creatine nitrate on muscle creatine content, body composition, anaerobic exercise capacity, bench press performance and clinical chemistry panels in recreationally active males.

ELIGIBILITY:
Inclusion Criteria:

* participants are apparently healthy and recreationally active males between the ages of 18 and 40;
* participants will need to have at least six months immediate prior history of resistance training on the bench press and leg press or squat;

Exclusion Criteria:

* participants have a history of treatment for metabolic disease (i.e., diabetes), hypertension, hypotension, thyroid disease, arrhythmias and/or cardiovascular disease;
* participants are currently using prescription medications;
* participants have a history of smoking;
* participants drink excessively (i.e., 12 drinks per week or more);
* participants have a recent history of creatine supplementation within six weeks of the start of supplementation;

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Effects of 28 Days of Different Forms of Creatine Supplementation on Body Water | 28 Days
  Assessing Body Water through Bioelectrical Impedance Analysis (BIA)
Effects of 28 Days of Different Forms of Creatine Supplementation on Body Composition | 28 Days
  Assessing Body Compositing through Dual-Energy X-Ray Absorptiometry (DXA)
Effects of 28 Days of Different Forms of Creatine Supplementation on intramuscular creatine | 28 Days
  Assessing intramuscular creatine using standard spectrophotometric methods using a microplate spectrophotometer
Effects of 28 Days of Different Forms of Creatine Supplementation on intramuscular phosphocreatine | 28 Days
  Assessing intramuscular phosphocreatine using standard spectrophotometric methods using a microplate spectrophotometer
Effects of 28 Days of Different Forms of Creatine Supplementation on intramuscular ATP | 28 Days
  Assessing intramuscular Adenosine Triphosphate (ATP) using standard spectrophotometric methods using a microplate spectrophotometer
Effects of 28 Days of Different Forms of Creatine Supplementation on muscular strength | 28 Days
  Assessing muscular strength through 1 Repetition Maximum (RM) testing
Effects of 28 Days of Different Forms of Creatine Supplementation on muscular endurance | 28 Days
  Assessing muscular endurance through repetition to failure testing
Effects of 28 Days of Different Forms of Creatine Supplementation on anaerobic capacity | 28 Days
  Assessing anaerobic capacity through 6 x 6 second sprints followed by a 30 second sprint on a Wingate bicycle ergometer

SECONDARY OUTCOMES:
Effects of 28 Days of Different Forms of Creatine Supplementation on training volume (weight lifted x number of repetitions x number of sets) | 28 Days
  Assessing training volume using a calculator
Effects of 28 Days of Different Forms of Creatine Supplementation on self-reported side effects | 28 Days
  Assessing self-reported side effects using a side effects questionnaire
Effects of 28 Days of Different Forms of Creatine Supplementation on blood | 28 Days
  Measure standard clinical chemistry panels in the blood to evaluate safety

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Kreider, PhD, Principal Investigator — Texas A&M University

IPD SHARING:
Plan to Share IPD: No